CLINICAL TRIAL: NCT04004507
Title: Single Dose Study of Phentolamine Mesylate Eye Drops in Patients With Severe Night Vision Disturbances
Acronym: SNV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ocuphire Pharma, Inc. (Industry)
Collaborators: Ophthalmic Consultants of Long Island (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NYX-SNV
Record Dates: First submitted 2019-06-28; First posted 2019-07-02 (Actual); Results first posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2022-05

CONDITIONS: Decrease in Night Vision; Disturbance; Vision, Loss
Keywords: Night Vision Disturbances; NVD; Glare; Halos; Starbursts; Nyxol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phentolamine Mesylate Ophthalmic Solution 1% (Experimental): 1 drop in each eye (QD) for one day.
  Interventions: Drug: Phentolamine Mesylate Ophthalmic Solution 1%
- Phentolamine Mesylate Ophthalmic Solution Vehicle (Placebo Comparator): 1 drop in each eye (QD) for one day.
  Interventions: Other: Phentolamine Mesylate Ophthalmic Solution Vehicle (Placebo)

INTERVENTIONS:
Drug: Phentolamine Mesylate Ophthalmic Solution 1% — Topical Sterile Ophthalmic Solution
  Arms: Phentolamine Mesylate Ophthalmic Solution 1%
Other: Phentolamine Mesylate Ophthalmic Solution Vehicle (Placebo) — Topical Sterile Ophthalmic Solution
  Arms: Phentolamine Mesylate Ophthalmic Solution Vehicle

SUMMARY:
The objectives of this study are:

* To assess the effect of ophthalmic phentolamine mesylate in mesopic conditions on the four endpoints:

  1. Contrast sensitivity
  2. Low contrast visual acuity
  3. Wavefront aberrometry
  4. Subjective questionnaire
* To assess the safety of ophthalmic phentolamine mesylate

DETAILED DESCRIPTION:
Double-masked, placebo-controlled, single-dose Phase 2 study in 24 patients experiencing severe night vision difficulties to evaluate ocular and systemic safety and efficacy following administration of one drop of phentolamine mesylate 1.0% QD in each eye for 1 day.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years of age
2. Currently experiencing severe night vision difficulty as reported subjectively
3. At least two patches below the normal range at any two frequencies in Contrast Sensitivity done under mesopic conditions with glare
4. Improvement in low contrast visual acuity (LCVA) in dim light during illumination of contralateral eye
5. Good general health
6. Written informed consent to participate in this trial
7. Ability to comply with all protocol mandated procedures and to attend all scheduled office visits

Exclusion Criteria:

1. Patients with untreated cataracts grades 1-4
2. Patients who wear contact lenses
3. Less than 5 weeks post-refractive surgery (LASIK or PRK)
4. Less than 5 weeks post intraocular lens insertion
5. Low blood pressure (systolic <120 mm Hg or diastolic <80 mm Hg)
6. A history of heart rate abnormalities
7. Administration of any investigational drug within 30 days of study initiation
8. Use of any eye drops with a pharmacologic effect on the pupil within 7 days of Visit 1
9. Use of any systemic alpha adrenergic antagonists (Appendix 1)
10. Known local or systemic hypersensitivity to adrenergic antagonists
11. For women of childbearing potential: currently pregnant or lactating, or unwilling to use birth control during the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-08 (Actual); Primary Completion 2007-10 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marguerite McDonald, MD, FACS, Principal Investigator — Ophthalmic Consultants of Long Island, NY
Locations (1):
- Ophthalmic Consultants of Long Island, NY, Lynbrook, New York, United States

REFERENCES:
- [Derived] Pepose J, Brigell M, Lazar E, Heisel C, Yousif J, Rahmani K, Kolli A, Hwang M, Mitrano C, Lazar A, Charizanis K, Sooch M, McDonald M. A randomized phase 2 clinical trial of phentolamine mesylate eye drops in patients with severe night vision disturbances. BMC Ophthalmol. 2022 Oct 8;22(1):402. doi: 10.1186/s12886-022-02621-6. PMID 36209072

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24 subjects were enrolled. Both eyes were treated and evaluated for efficay and safety.
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | Phentolamine Mesylate Ophthalmic Solution 1% | Phentolamine Mesylate Ophthalmic Solution Vehicle
Started | 16; 32 eyes | 8; 16 eyes
Completed | 16; 32 eyes | 8; 16 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: 24 subjects were enrolled. Both eyes were evaluated for efficacy and safety.
Units Other Than Participants: eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | Phentolamine Mesylate Ophthalmic Solution 1% | Phentolamine Mesylate Ophthalmic Solution Vehicle | Total
Number analyzed (Participants) | 16 | 8 | 24
Number analyzed (eyes) | 32 | 16 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (14.6) | 47.4 (13.5) | 43.9 (19.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 5 | 17
  Male | 4 | 3 | 7
Pupil Diameter Illuminated [Mean (Standard Deviation); unit: mm] | 4.4 (0.6) | 4.9 (0.8) | 4.6 (1)
Trans-Illuminated Low Contrast Visual Acuity [Mean (Standard Deviation); unit: Letters] | 33.1 (5.4) | 30.1 (8.4) | 32.1 (10.0)

OUTCOME MEASURES:

1. Primary Outcome: Contrast Sensitivity
Description: Average change in monocular contrast sensitivity scores under mesopic conditions at each of five spatial frequencies with and without glare.
  The tests were performed in a darkened room using the Optec 6500 instrument (Stereo Optical) using Slides 5-9 (spatial frequencies 1.5 - 18 cycles per degree), with the distance setting at "far", and with the light setting at "night". Subjects were asked to read each slide from left to right indicating if the lines were tilted to the left, the right or straight up and down until they provided 2 consecutive incorrect responses. The total number of correct responses for each slide was recorded.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Patches
Units Other Than Participants: Eyes
Arm/Group | Phentolamine Mesylate Ophthalmic Solution 1% | Phentolamine Mesylate Ophthalmic Solution Vehicle
Number analyzed (Participants) | 16 | 8
Number analyzed (Eyes) | 32 | 16
Patches
  1.5 Cycles with Glare | 0.6 (1.8) | 0.8 (1.5)
  3 Cycles with Glare | 0.9 (2.1) | 0.7 (1.5)
  6 Cycles with Glare | 1.4 (1.9) | 0.1 (1.3)
  12 Cycles with Glare | 1.7 (2.0) | 0.4 (1.0)
  18 Cycles with Glare | 1.3 (1.8) | 0.3 (0.8)
  1.5 Cycles without Glare | 1.0 (1.4) | 0.4 (1.4)
  3 Cycles without Glare | 1.3 (1.5) | 0.7 (1.3)
  6 Cycles without Glare | 1.1 (1.4) | 0.5 (1.4)
  12 Cycles without Glare | 0.8 (1.6) | -0.2 (1.0)
  18 Cycles without Glare | 0.5 (1.4) | 0.3 (0.9)

2. Secondary Outcome: Visual Acuity
Description: Average number of letters of improvement in the following parameters:
  1. Distance high-contrast visual acuity under mesopic conditions (monocular, measured at 4 meters)
  2. Distance high-contrast visual acuity under photopic conditions (monocular, measured at 4 meters)
  3. Distance low-contrast visual acuity under mesopic conditions (monocular, measured at 4 meters)
  4. Distance low-contrast visual acuity under photopic conditions (monocular, measured at 4 meters)
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Letters
Units Other Than Participants: Eyes
Arm/Group | Phentolamine Mesylate Ophthalmic Solution 1% | Phentolamine Mesylate Ophthalmic Solution Vehicle
Number analyzed (Participants) | 16 | 8
Number analyzed (Eyes) | 32 | 16
Letters
  Distance high-contrast visual acuity under mesopic conditions | 6.5 (7.2) | 1.1 (3.9)
  Distance high-contrast visual acuity under photopic conditions | 3.8 (7.6) | 0.1 (3.8)
  Distance low-contrast visual acuity under mesopic conditions | 8.0 (8.4) | 3.1 (4.5)
  Distance low-contrast visual acuity under photopic conditions | 7.3 (6.6) | 0.9 (3.6)

3. Secondary Outcome: Self-Reported Vision Quality
Description: Subjective patient evaluations of vision quality at night (% rating their vision as improved)
Time Frame: 1 day
Measure: Number; unit: Percentage
Arm/Group | Phentolamine Mesylate Ophthalmic Solution 1% | Phentolamine Mesylate Ophthalmic Solution Vehicle
Number analyzed (Participants) | 16 | 8
Percentage | 69 | 75

4. Secondary Outcome: Pupil Diameter
Description: Average change in pupil diameter
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Eyes
Arm/Group | Phentolamine Mesylate Ophthalmic Solution 1% | Phentolamine Mesylate Ophthalmic Solution Vehicle
Number analyzed (Participants) | 16 | 8
Number analyzed (Eyes) | 32 | 16
mm | -1.3 (0.8) | -0.2 (0.5)

ADVERSE EVENTS:
Arm/Group | Phentolamine Mesylate Ophthalmic Solution 1% | Phentolamine Mesylate Ophthalmic Solution Vehicle
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/8
Other Adverse Events (participants affected / at risk) | 0/16 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No